CLINICAL TRIAL: NCT03727685
Title: Multi-channel Dissemination of Information for Digital Advance Care Planning Platform (Our Care Wishes) to Hospital Admits
Brief Title: Disseminating a Digital ACP Platform (Our Care Wishes) to Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Scott Halpern, Professor of Medicine, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 831901
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Hospitalism
Keywords: Advance care planning

STUDY DESIGN:
Intervention Model Description: The design is a stepped-wedge cluster design in which specific areas of the hospital will adopt the intervention, in sequence. All areas of the hospital will begin in the control phase. 12 weeks into the study period, the first "wedge" or area of the hospital will adopt the Our Care Wishes intervention, 4 weeks after, the next wedge will switch the control phase, the final wedge will adopt the intervention after that.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Patients admitted to the hospital will not receive information about Our Care Wishes.
- Intervention: Our Care Wishes (Active Comparator): Patients admitted to the hospital during the intervention phase will receive information from registration representatives regarding Our Care Wishes.
  Interventions: Behavioral: Our Care Wishes

INTERVENTIONS:
Behavioral: Our Care Wishes — A flyer describing the Our Care Wishes platform will be added to the back pocket of admission packets for patients being admitted via the Silverstein 1 Admission Office and the Emergency Department and for patients being seen in the Pre Admission Testing office. Registration reps in these locations will inform all patients seen that Penn has created a free, online resource called Our Care Wishes to help patients with Advance Care Planning and ask if they would like to be sent a link to Our Care Wishes by email or text. For those patients who respond affirmatively, the rep will then complete the necessary fields to refer on www.ourcarewishes.org/refer.
  Arms: Intervention: Our Care Wishes

SUMMARY:
Penn Medicine has created a novel, online, evidence-based advance care planning (ACP) platform through its Center for Health Care Innovation. The platform is called "Our Care Wishes" and utilizes a 'shopping-cart' approach to ACP, allowing users to name surrogate decision makers, make choices about quality of life and medical treatments, outline medical wishes and organ donation, and share preferences for their end of life experience. Our Care Wishes then creates an easy to read, updatable ACP document that can be electronically shared with loved ones and uploaded to a patient's electronic medical record in PennChart.

It is believed that this platform may help to overcome engagement and infrastructure barriers previously identified in the literature regarding the completion of ACP documents. The intervention will consist of multi-channel information dissemination regarding Our Care Wishes to Hospital of the University of Pennsylvania patients admitted through two locations (the Emergency Department, Silverstein 1 Admission Office) and outpatients who are seen in Pre-Admission Testing (PAT). All patients visiting these two locations during the intervention phase will receive a paper handout with information regarding Our Care Wishes included in their customary admission folder packet. The registration representative (RR) at these three locations will provide a brief explanation of the site as they check the patients in, as well send the patients a direct link to the site for non-ED admits via email and text message.

DETAILED DESCRIPTION:
Registration representatives (RR) from Silverstein 1 Admission Office, the Emergency Department, and the Pre Admission Testing office will be administering the intervention at the three sites. The current workflow is for the RR to provide all new admits with an admission packet created by Guest Services and also ask ALL patients whether they have completed an Advance Directive as mandated by the Patient Self-Determination Act of 1991 with little attention paid to encouraging AD completion. During the control/baseline phase of this trial, this workflow will remain the same.

During the intervention phase, a flyer describing the Our Care Wishes platform will be added to the back pocket of admission packets for patients being admitted via the Silverstein 1 Admission Office and the Emergency Department and for patients being seen in the Pre Admission Testing office. The interventions will vary slightly between Silverstein 1/PAT and the Emergency Department given concern for limited bandwidth by RR in the ED setting.

For patients admitted through Silverstein 1 and who visit PAT, they will present to the RR per usual and the RR will follow the current workflow. At the point where the RR asks the patient if they have an AD and if it is present, the RR will remind the patient of the importance of having a document that records their care wishes. The RR will then inform the patient that Penn has created a free, online resource called Our Care Wishes to help patients with Advance Care Planning. The platform allows patients to upload their wishes right into PennChart using their MyPennMedicine login. The RR will then show the flyer in the back pocket of the admission folder to the patient. For patients being admitted via Silverstein 1 Admission Office and those being seen in the Pre Admission Testing office, the RR will then proceed to ask patients if they would like to be sent a link to Our Care Wishes by email or text. For those patients who respond affirmatively, the RR will ask for the preferred email or phone number and will then complete the necessary fields to refer on www.ourcarewishes.org/refer.

For patients admitted through the Emergency Department, a weekly report will be created that generates a list of admissions during the prior week along with their active PennChart email address and date of death if applicable (maternal and child health will be excluded). The research coordinator will email non-deceased patients 7-14 days after their admission date. The email will be sent to patients with an email address in PennChart. The email will not include any personally identifiable information regarding the patient or mention of their recent admission/visit. The email will include high-level information regarding Our Care Wishes, effectively summarizing the information that the patient received in their admission folder and stating the value of ACP, along with a direct link to access Our Care Wishes.

For this process, it is estimated that the RR will spend 60-90 seconds noting the presence of the handout in the admissions folder and sending the patient a direct link (for those that opt-in). Frequency of the intervention will be every patient admitted via Silverstein 1 Admissions office and seen in Pre-Admission Testing during the intervention timeframe.

Each week, a report will be constructed via EPIC reporting to identify the patients that are admitted via these offices during this timeframe. The report will be made available to only key personnel on this research study. The report will also include this information which is routinely collected during the course of a hospitalization:

* Demographics (date of birth, sex, etc.)
* Date of death (if recorded in the EHR)
* Place of death (if recorded in the EHR)
* Dates of hospitalization(s)
* Contact information (email address and mobile phone number)MRN
* HAR
* Name
* Unit admitted to
* Presence of AD in EHR
* Admission source (need ED and Silver 1)
* Outside hospital transfer? (exclude if yes)
* Mother/baby? (exclude if yes)
* PAT appointment date

ELIGIBILITY:
Inclusion Criteria:

* Adult admitted at the University of Pennsylvania via two locations: the Emergency Department, Silverstein 1 admission office;
* Patients that are seen in the Pre-Admission Testing (PAT) clinic
* Patients must speak English fluently

Exclusion Criteria:

* Maternity patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16020 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
New Presence of ACP | within two months of the index visit
  Presence of an uploaded advance care planning document that shares any care wishes or preferences (beyond simply naming a surrogate)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Halpern, Ph.D, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- See also: Main intervention — http://Ourcarewishes.org